CLINICAL TRIAL: NCT00784758
Title: Effect of Fenzian™ Treatment on Symptoms, Pulmonary Function and Albuterol/Salbutamol Use in Patients With Mild to Moderate Persistent Asthma: A Multicenter, Sham-Controlled Clinical Trial
Brief Title: Fenzian Asthma Multicenter Outcomes Study
Acronym: FAMOUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Fenzian Ltd. (Unknown)
Responsible Party: Principal Investigator, Eric Kleerup, Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Fenzian
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Asthma
Keywords: Asthma; Lung Diseases; Respiratory Tract Diseases
MeSH Terms: conditions — Asthma; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fenzian Device (Experimental): Subjects randomized to this arm will receive treatment with the Fenzian Device
  Interventions: Device: Fenzian Device
- Sham Device (Sham Comparator): Subjects randomized to this arm will receive treatment with the sham device.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Fenzian Device — Three 20-minute treatments with the Fenzian Device per week for 5 weeks (for a total of 15 treatments)
  Arms: Fenzian Device
Device: Sham Device — Three 20-minute treatments with the sham device per week for 5 weeks (for a total of 15 treatments) (NOTE: This arm is similar to a placebo arm in a drug trial.)
  Arms: Sham Device

SUMMARY:
The purpose of this study is to investigate the effects of Fenzian™ treatment on symptoms (such as shortness of breath), lung function (how well the lungs work), and albuterol/salbutamol (rescue medication) use in people with asthma. This will be done by comparing the effects of Fenzian™ treatment to the effects of a sham treatment, which looks the same as the Fenzian™ device but doesn't do anything.

The Fenzian™ device is an electrical instrument that the investigators hope will help reduce airway inflammation associated with asthma symptoms by stimulating the nerves with very low electrical currents. The study device will be applied directly to the skin on the back, working along the ribs toward the spine, alternating between left and right sides, and on your face.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-80 years. [NOTE: Only the Johns Hopkins site will enroll subjects under 18.]
* Clinical history consistent with asthma (GINA 4 definitions) for at least six months
* Current symptoms and features of partly-controlled or uncontrolled asthma, according to GINA classification of asthma control
* A stable (1 month) treatment regimen consisting of:

  * as needed short-acting bronchodilators alone,
  * as needed short-acting bronchodilators in combination with low- or medium-dose inhaled corticosteroids (<= 1000 mcg per day beclomethasone or equivalent,
  * any combination of long acting beta-agonist bronchodilator and low- or medium-dose inhaled corticosteroid (as defined above),as needed short-acting bronchodilators in combination with montelukast or other leukotriene modifier
* Willingness to comply with the study protocol and ability to perform the study procedures.
* Willingness to attend the study site according to the specified treatment schedule

Inclusion Criteria Assessed at Visit 1:

* Pre-bronchodilator forced expiratory volume at one second (FEV1) between 60% predicted and the lower limit of normal.
* Pre-bronchodilator [FEV1/forced vital capacity (FVC)] less than the lower limit of normal.
* Reversibility of FEV1 of at least 200 ml, 15-20 minutes after 4 puffs of albuterol HFA pressurized metered-dose inhaler pMDI.

Inclusion Criteria Assessed at Visit 2:

* Reversibility of FEV1 of at least 200ml, 15-30 minutes after 4 puffs of albuterol HFA pressurized metered-dose inhaler (pMDI) if not confirmed at Visit 1 plus
* Using short-acting bronchodilator therapy on two or more occasions in each of the two weeks preceding Visit 2 plus (Ventolin HFA counter decrease of at least 8 puffs)
* Partly controlled or uncontrolled of asthma as indicated by one to three, but not four of the following in each of the two weeks preceding Visit 2:

  * Daytime symptoms more than twice per week
  * Any limitation of activity
  * Any nocturnal symptoms or awakening
  * peak expiratory flow (PEF)<80% of predicted on any day

Exclusion Criteria:

* Pulmonary disease other than asthma, such as smoking-related chronic obstructive pulmonary disease (COPD), clinically significant bronchiectasis, lung resection, and interstitial lung disease.
* Other significant systemic illness which might, in the opinion of the investigator alter the risk or outcome of the study (e.g. cardiovascular arrhythmias or conduction abnormalities, hyperthyroidism, uncontrolled hypertension, cancer)
* Tobacco smoking greater than 10 pack-year of cumulative exposure or current smoking within 10 years.
* Respiratory tract infection within 6 weeks of the study.
* Seasonal allergies causing symptoms within the past 4 weeks. Perennial or out of season allergic rhinitis is acceptable. Nasal corticosteroids and long-acting antihistamines are acceptable.
* Any investigational drug or treatment within 30 days.
* Use of cromolyn, nedocromil, theophylline, tiotropium, or oral albuterol within 1 week prior to Visit 1 of the study.
* Current use of omalizumab or within the last 8 weeks.
* Subjects on anti-depressant (mono-amine oxidase inhibitors or tricyclic antidepressants) treatment within 8 weeks.
* Non-potassium sparing diuretics unless in fixed combination with potassium-sparing diuretics within one week.
* Digoxin, within one week, unless levels have been monitored previously while taking albuterol or long-acting beta2-agonist (LABAs).
* Presence of an implanted cardiac pacemaker or neurostimulator. A removable transcutaneous nerve stimulator, not used during the treatment sessions is acceptable.
* Non-selective beta agonists. (acceptable choices include: bisprolol, betaxolol, atenolol, acebutolol and metoprolol)
* Subjects who are pregnant or breast feeding.
* Persons employed by or related to those employed by the investigative site (e.g. Pulmonary Division).
* Prior Fenzian treatment for any indication
* Hypersensitivity or intolerance of albuterol HFA pMDI (Ventolin) or its components. Note: if the subject is using ipratropium bromide for rescue short-acting bronchodilator, they must specifically not have been placed on that treatment due to intolerance of albuterol/salbutamol.
* Inability to withhold, before and during each visit (except the initial consent visit), xanthine-containing foods (coffee, tea, cola, chocolate, etc.) and alcohol for 6 hours, and short-acting bronchodilators for 8 hours.
* Unwillingness to stop use of non-study supplied albuterol (nebulized, chlorofluorocarbon (CFC) or HFA), other short-acting beta agonists (e.g. epinephrine, levalbuterol, metaproterenol, pirbuterol, terbutaline) and ipratropium during the study (after consent through visit 4).
* Inability to coordinate the timing for doses of long-acting beta agonists (withhold period at least 12 hours prior to visit) with Visits 1, 2, 3 or 4

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B Cooper, M.D., Principal Investigator — University of California, Los Angeles
Locations (6):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
- University of Cape Town Lung Institute, Mowbray, Cape Town, South Africa
- United Kingdom (2):
  - Addenbrookes NHS Trust, Cambridge University, Bottisham, Cambridgeshire
  - London Chest Hospital, London, England

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at six clinical sites using flyers, newspaper, radio and campus advertising, and by contacting participants of prior studies whom agreed to future contacts. The recruitment period lasted from June 2009 to December 17, 2010.
Pre-assignment Details: Participants who signed consent and passed screening were enrolled into the study and randomized to a treatment arm. One of 42 active treatment participants withdrew consent after being randomized but prior to receiving treatment. He/she did not provide a reason.
Groups:
- Fenzian Device: 20-minute treatments with the Fenzian Device, 3 times per week for 5 weeks (15 treatments total)
- Sham Device: 20-minute treatments with the sham device, 3 times per week for 5 weeks (15 treatments total).
Period: Overall Study
Arm/Group | Fenzian Device | Sham Device
Started | 42 | 39
Began Treatment | 41 | 39
Completed Treatment | 40 | 39
Completed | 38 | 39
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fenzian Device | Sham Device | Total
Number analyzed (Participants) | 42 | 39 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 39 | 80
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (13.1) | 37.2 (13.4) | 37.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 21 | 23 | 44
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
  South Africa | 26 | 22 | 48
  United Kingdom | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Asthma Control Questionnaire (ACQ) 7 Score
Description: Asthma Control Questionnaire (QOL Technologies 2004) Elizabeth Juniper, (Eur Respir J 1999; 14:902-7). Range 0-6, 0 is no symptoms, 6 is maximal symptoms. 0.5 is considered a minimally important difference, 0.75 or less is associated with a 85% chance that the subject's asthma is well controlled, 1.50 or greater is associated with a 88% chance that the subject's asthma is not well controlled. The ACQ consists of 6 patient/subject reported questions on symptoms and a question completed by the staff for categorization of the patient/subjects forced expiratory volume in the first second (FEV1) from spirometry.
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed Visit 3 (5 weeks of treatment) were included in the analysis.
Measure: Mean (Standard Error); unit: ACQ7 score
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
ACQ7 score | -0.35 (0.08) | -0.29 (0.08)

2. Secondary Outcome: Daily Short-acting Bronchodilator (Albuterol/Salbutamol) Use
Description: Daily short-acting bronchodilator use during the 2 weeks, modeled as a zero-modified negative binomial (usually 2 puffs/day)
Time Frame: 2 weeks after completion of treatment (weeks 9-11)
Population: All subjects whose short-acting bronchodilator counters were functioning and who completed Visit 3 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Puffs/day
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 28 | 29
Puffs/day | 0.83 (1.58) | 0.71 (1.23)

3. Secondary Outcome: Short-acting Bronchodilator (Albuterol/Salbutamol) Free Days
Description: Percent of rescue-free days during a two week period after completing treatment phase
Time Frame: 2 weeks after completion of treatment (weeks 10 -11)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percent of days
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 28 | 24
Percent of days | 63 [45 to 81] | 60 [40 to 60]

4. Secondary Outcome: Change in Asthma Control Questionnaire 6 Score
Description: Asthma Control Questionnaire (QOL Technologies 2004) Elizabeth Juniper, (Eur Respir J 1999; 14:902-7). Range 0-6, 0 is no symptoms, 6 is maximal symptoms. 0.5 is considered a minimally important difference, 0.75 or less is associated with a 85% chance that the subject's asthma is well controlled, 1.50 or greater is associated with a 88% chance that the subject's asthma is not well controlled. The ACQ consists of 6 patient/subject reported questions on symptoms.
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed Visit 3 were included in the analysis.
Measure: Mean (Standard Error); unit: ACQ6 score
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
ACQ6 score | -0.40 (0.09) | -0.29 (0.09)

5. Secondary Outcome: Change in Spirometry - FEV1
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed Visit 3 were included in the analysis.
Measure: Mean (Standard Error); unit: L
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
L | 0.00 (0.04) | 0.09 (0.04)

6. Secondary Outcome: Change in Spirometry - Forced Vital Capacity (FVC)
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed Visit 3 were included in the analysis.
Measure: Mean (Standard Error); unit: L
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
L | -0.07 (0.04) | 0.04 (0.04)

7. Secondary Outcome: Change in Spirometry - FEV1/FVC
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed Visit 3 were included in the analysis.
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
Ratio | 0.81 (1.14) | 1.97 (1.13)

8. Secondary Outcome: Change in Spirometry FEF25-75%
Description: A measure of forced expiratory flow between 25% and 75% of FVC (FEF25-75%)
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed treatment (weeks 5-9) were included in the analysis.
Measure: Mean (Standard Error); unit: L/s
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
L/s | 0.01 (0.07) | 0.19 (0.06)

9. Secondary Outcome: Change in Asthma Control Test Score
Description: The Asthma Control Test is a 5-item questionnaire using 1-5 point Likert scales; maximum score 25 = complete control of asthma; minimum score 5 = poor control of asthma.
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed Visit 3 were included in the analysis.
Measure: Mean (Standard Error); unit: ACT score
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
ACT score | 1.49 (0.37) | 0.69 (0.37)

10. Secondary Outcome: Change in Mini Asthma Quality of Life Questionnaire (AQLQ) Score (to Evaluate Quality of Life)
Description: The mini AQLQ is a questionnaire specifically designed to assess health status in patients with asthma. The mini-AQLQ consists of 15 questions covering symptoms and activities. Each question is scaled from 1 (poorly controlled asthma) to 7(maximally controlled asthma) where 7 reflects a higher quality of life. Total score is the sum of 15 items and may range from 15-105. An increase in the AQLQ score indicates a better quality of life.
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed Visit 3 were included in the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
units on a scale | 0.56 (0.99) | 0.31 (0.10)

11. Secondary Outcome: Change in Sino-Nasal Outcome Test (SNOT-22) - Total Score
Description: The SNOT-22 is a disease-specific quality of life score for rhinosinusitis. SNOT22 is a validated scale which measures sinonasal symptoms for sinusitis patients. The 22 questions are rated on a scale of 0-5 for a maximum total score of 110. Higher scores represent more symptomatic patients.
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed Visit 3 were included in the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
units on a scale | 0.74 (0.31) | 0.02 (0.34)

12. Secondary Outcome: Change in SNOT-22 Nasal Sub-score
Description: Sino-nasal outcome test-22 nasal sub-score. The nasal subscore consists of 8 questions, each on a scale of 0 (no problems) to 5 (as bad as it can be). Higher scores indicate worse symptoms of rhinosinusitis.
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed Visit 3 were included in the analysis.
Measure: Mean (Standard Error); unit: SNOT22 score
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
SNOT22 score | 0.26 (0.37) | 0.23 (0.40)

13. Secondary Outcome: Daytime Symptom Score
Description: Daytime symptoms due to asthma were assessed via the electronic diary (AM2+ Asthma Monitor) each evening for 7 days prior to the study visit at Week 15. Daily scores were derived from five questions relating to 1) frequency of asthma symptoms, 2) impact of asthma symptoms, 3) activity, 4) impact of asthma on activity, and 5) breathlessness. Each question was scored from 0 (best) to 6 (worst), with the average of 5 questions providing a daily score ranging from 0 (best) to 6 (worst). Each participant's symptom score was calculated as the average of 7 daily scores. Thus, the range of possible scores is from 0 (best) to 6 (worst).
Time Frame: 7 days prior to final assessment visit at week 15
Population: All subjects whose diaries were functioning and who completed diary assessments and completed Visit 3 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 13 | 14
score on a scale | 0.83 (0.81) | 0.65 (0.58)

14. Secondary Outcome: Change in Transition Dyspnea Index (TDI) - Functional Impairment
Description: The TDI is an interviewer-administered instrument which measures the changes in the participant's dyspnea from Baseline. The scores in the TDI evaluate ratings for 3 different categories (functional impairment, magnitude of task in exertional capacity, and magnitude of effort). TDI category scores range from -3 (major deterioration) to +3 (major improvement)
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed Visit 3 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
units on a scale | 0.87 (1.00) | 0.25 (0.69)

15. Secondary Outcome: Change in Transition Dyspnea Index - Magnitude of Task at Visit 3
Description: as for outcome 14
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed Visit 3 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
units on a scale | 0.84 (0.92) | 0.34 (0.76)

16. Secondary Outcome: Change in Transition Dyspnea Index - Magnitude of Effort at Visit 3
Description: as for outcome 14
Time Frame: Baseline to completion of treatment at 9 weeks
Population: All subjects who completed Visit 3 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 40 | 39
units on a scale | 0.87 (0.96) | 0.40 (0.95)

17. Secondary Outcome: Change in Transition Dyspnea Index - Functional Impairment
Description: as for outcome 14
Time Frame: Baseline to final assessment visit (15 weeks)
Population: All subjects who completed Visit 4 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 38 | 39
units on a scale | 0.72 (1.10) | 0.41 (1.00)

18. Secondary Outcome: Change in Transition Dyspnea Index - Magnitude of Task
Description: as for outcome 14
Time Frame: Baseline to final assessment visit (15 weeks)
Population: All subjects who completed Visit 4 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 38 | 39
units on a scale | 0.62 (1.00) | 0.43 (1.10)

19. Secondary Outcome: Change in Transition Dyspnea Index - Magnitude of Effort
Description: as for outcome 14
Time Frame: Baseline to final assessment visit (15 weeks)
Population: All subjects who completed Visit 4 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fenzian Device | Sham Device
Number analyzed (Participants) | 38 | 39
units on a scale | 0.69 (1.10) | 0.41 (1.10)

ADVERSE EVENTS:
Time Frame: 15 weeks for each subject
Description: All reported adverse events, regardless of relatedness to study
Arm/Group | Fenzian Device | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 28/40 | 21/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fenzian Device (N=40) | Sham Device (N=39)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 | 3 — Worsening of asthma
Other dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper respiratory infections (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Other infection (Infections and infestations) | 4 | 1 — One of each of the following: Conjunctivitis, Infected scalp lesion, fungal fingernail infection, Otitis media (ear infection), urinary tract infection
Candidiasis, Oral (Infections and infestations) | 1 | 1
Exanthema (Skin and subcutaneous tissue disorders) | 2 | 1 — Skin rash
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Injury (Injury, poisoning and procedural complications) | 1 | 1
Sweating (Skin and subcutaneous tissue disorders) | 3 | 1
Edema (Skin and subcutaneous tissue disorders) | 0 | 1 — Pedal edema
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diabetes Mellitus, Type 2 (Endocrine disorders) | 1 | 0
Weight loss (General disorders) | 1 | 0
Central Nervous System Disorders (Nervous system disorders) | 3 | 0 — Dizziness, anxiety, headache
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — Lower respiratory tract infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The University (the PI) must furnish the Sponsor with a copy of any proposed written or oral publication (including manuscripts, abstracts, and oral presentations) at least 30 days prior to submission for publication. The Sponsor can direct the PI to delete their confidential information. The information contained in this results section was provided to the Sponsor 30 days ago and they have not asked for any deletions.